CLINICAL TRIAL: NCT07372495
Title: Cervical Cerclage Plus Vaginal Progesterone Versus Vaginal Progesterone Alone in Twin Pregnancies With a Short Cervix for Prevention of Preterm Birth: a Randomized Controlled Trial
Brief Title: Cerclage Plus Progesterone vs Progesterone Alone in Twin Short Cervix
Acronym: VNTWINC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital of Obstetrics and Gynecology (Other)
Collaborators: Quang Ninh Obstetrics and Pediatrics Hospital, Quang Ninh, Vietnam (Other); Ninh Binh Obstetrics and Pediatrics Hospital, Ninh Binh, Vietnam (Other); Bac Ninh 1 Obstetrics and Pediatrics Hospital, Bac Ninh, Vietnam (Unknown); Bac Ninh 2 Obstetrics and Pediatrics Hospital, Bac Ninh, Vietnam (Unknown); Hung Yen Obstetrics and Pediatrics Hospital, Hung Yen, Vietnam (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHOG-VN.TWIN CERCLAGE
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Preterm
Keywords: Twin pregnancy; cervical cerclage; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical; Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either cerclage plus progesterone or progesterone alone in a 1:1 ratio with a variable block size of 4 or 6.
Masking Description: Participants and investigators will not be blinded for the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerclage plus progesterone (Experimental): Participants will receive cervical cerclage according to local protocols within one week after randomization. The procedure will be performed by three senior clinicians experienced in cerclage, using the McDonald technique. In addition, vaginal micronized progesterone will be administered at a total daily dose of 400 mg, given as Utrogestan® 200 mg (Besins Healthcare, France) twice daily, in the morning and at bedtime. Participants will be asked to record their vaginal progesterone application in a patient diary sheet for up to 140 days.
  Interventions: Procedure: Cervical cerclage; Drug: Progesterone
- Progesterone alone (Active Comparator): Vaginal micronized progesterone will be administered at a total daily dose of 400 mg, given as Utrogestan® 200 mg (Besins Healthcare, France) twice daily, in the morning and at bedtime. Participants will be asked to record their vaginal progesterone application in a patient diary sheet for up to 140 days
  Interventions: Drug: Progesterone

INTERVENTIONS:
Procedure: Cervical cerclage — Participants will receive cervical cerclage according to local protocols within one week after randomization. The procedure will be performed by two to three senior clinicians experienced in cerclage in each center, using the McDonald technique.
  Arms: Cerclage plus progesterone
Drug: Progesterone — Vaginal micronized progesterone will be administered at a total daily dose of 400 mg, given as Utrogestan® 200 mg (Besins Healthcare, France) twice daily, in the morning and at bedtime. Participants will be asked to record their vaginal progesterone application in a patient diary sheet for up to 140 days.
  Other Names: Utrogestan 200mg

SUMMARY:
This study aims to compare the effectiveness of cervical cerclage combined with progesterone versus progesterone alone in preventing preterm birth among women with twin pregnancies and a short cervix (cervical length ≤ 30 mm). Participants will be randomly allocated to either the intervention group (cerclage plus progesterone) or the control group (progesterone alone).

DETAILED DESCRIPTION:
The incidence of multiple pregnancies has increased rapidly over the years mainly due to the resultant widespread use of assisted reproduction techniques. The twin birth rate in the USA has risen 70%, from 19 per 1000 live births in 1980 to 31 per 1000 live births in 2020. Twin pregnancies have a high risk on preterm birth (PTB) which is associated with increased risk of neonatal mortality and long-term morbidity. Around 60% of twin pregnancies deliver prior to 37 weeks and 12% before 34 weeks of gestation, with rates 5 and 8 times higher than the equivalent rates for a singleton pregnancy, respectively. Children born at an early gestational age are at increased risk of short-term morbidities affecting vital organ systems such as lungs, brain, bowels and are at increased risk of severe infection and sepsis. Perinatal mortality is strongly associated with extreme PTB. Survivors are at increased risk for developmental and behavioral disorders. In Vietnam, the rate of twin pregnancies deliver at < 28 weeks was about 11% in 2019. Caring for extremely premature infants is a significant burden for families and society. Therefore, obstetricians have a need for high-quality evidence for effective treatments.

Cervical length measurement (ideally transvaginal) is the preferred method of screening for preterm birth in twins; 25mm is a pragmatic cut-off between 18 and 24 gestational weeks (Grade of recommendation: C). Majority of the studies conducted previously has taken the cut-off cervical length as ≤ 25 mm. A systematic review and meta-analysis (13 retrospective studies and 3 RCTs) showed that cervical cerclage may reduce preterm birth in twin pregnancies with a cervical length <25 mm; however, preterm birth before 37, 34, and 28 weeks remained high (56.7%, 38.8%, and 11.7%, respectively)5, compared with much lower rates in singleton pregnancies (6.2%, 4.7%, and 0.4%). These findings support the need for further studies on preterm birth prevention in twin pregnancies with a cervical length >25 mm. In 2025, Yen et al. showed that cervical cerclage was more effective than pessary in twin pregnancies with a cervical length ≤28 mm, particularly in reducing preterm birth <28 weeks, with benefit observed at 25-28 mm. However, preterm birth rates remained high, suggesting that intervention at a higher cervical length threshold may be justified. Given gestational age-related cervical shortening and the substantially higher preterm birth risk in twins, a higher threshold corresponding to the 10th percentile (≤30 mm) has been proposed. Accordingly, we selected ≤30 mm as the intervention threshold in twin pregnancies.

In singleton pregnancies, vaginal progesterone is recommended as the primary intervention for pregnant women with a cervical length less than 25mm with consistently demonstrated effectiveness in preventing premature labor. In cases with a prior spontaneous preterm delivery and a short cervix, the placement of a vaginal cerclage should be considered. Conversely, there is less evidence on the optimal strategy for preventing PTB in twin pregnancies. In twins, IM 17- OHPC and cervical pessary are not indicated in order to prevent PTB. Evidence regarding the effectiveness of vaginal progesterone and cerclage remains unclear. Several randomized trials and systematic reviews reported little or no benefit of cerclage in twin pregnancies. However, these studies were limited by small sample size and large heterogeneity in their inclusion criteria, study populations, and outcomes observed. The data are insufficient to recommend for or against these interventions in the clinical circumstances. Moreover, in the a last few years, an increasing number of studies reporting a potential beneficial role of cerclage in reducing the risk of PTB and adverse outcomes in twin pregnancies have been published. The latest ISUOG practice guidelines (2025) stated that a combined strategy of physical-exam-indicated cerclage, antibiotics, and tocolytics may be considered in asymptomatic twin pregnancy with dilated cervix before 24 weeks of gestation and a cervical cerclage may be considered when the cervical length is ≤ 15 mm before 24 weeks of gestation (grade of recommendation: C). However, these findings are mainly based on observational studies and require confirmation in large and adequately powered RCTs.

In conclusion, there is a lack of well-designed RCT's on the effect of vaginal cerclage in asymptomatic twin pregnancies. We propose a multi-center randomized trial on the effectiveness of vaginal cerclage in women with a twin pregnancy and a short cervix (less than 30mm) in the second trimester with relevant outcomes assessing not only PTB at different cut-offs but also adverse maternal and neonatal outcomes.

This open label, multi-center, randomized controlled trial aims to compare the effectiveness of cervical cerclage combined with progesterone versus progesterone alone in preventing preterm birth among women with twin pregnancies with a cervix ≤ 30 mm.

Cervical length will be measured routinely in twin pregnancies between 16 and 24 weeks of gestation by qualified doctors via transvaginal ultrasound. Women with a cervical length ≤30 mm will be eligible for the study. Eligible participants will receive a Participant Information Sheet and provide written informed consent after discussion with the investigators. All eligible women will be invited to participate in the study.

Six centers are involved in the study and patients will be stratified by center. Patients will be randomly assigned in a 1:1 ratio to receive either cerclage plus progesterone or progesterone alone, using block randomization with a variable block size of 4, 6. To ensure allocation concealment, the random lists will be generated by www.sealedenvelope.com. Upon identification of an eligible participant, randomization data will be sequentially accessed an administrative staff who does not involve in clinical intervention. The random allocation will be conveyed to responsible clinicians. Due to the nature of interventions, the obstetricians and patients will not be blinded. Apart from randomization, patients will be managed and treated preterm birth (if present) according to local protocol.

In participants allocated to cerclage plus progesterone group, a Mersilene suture (Ethicon, LLC, United State) will be placed around the cervix in a purse-string fashion and securely tied anteriorly, following the McDonald technique under spinal anesthesia. The intervention needs to be performed before 24+0 weeks of gestation, by a team of dedicated obstetricians in our hospitals (2 to 3 obstetricians in each centers) to ensure the quality of the surgical procedure. For standardization of the cervical cerclage technique, all participating physicians received standardized training before study initiation. Prophylactic antibiotic: First/Second - generation Cephalosporin will be administered intravenously 1 hour before the procedure. In case of reporting an allergy to Cephalosporin, Clindamycin (Dalacin C® 600mg/4ml Pfizer, Belgium) will be used. Additional vaginal micronized progesterone will be administered at a total daily dose of 400 mg, given as Utrogestan® 200 mg (Besins Healthcare, France) twice daily, in the morning and at bedtime, from 2 days after receiving cerclage to 37+0/7 week of gestation or preterm birth whatever comes first.

In participants allocated to progesterone alone group, vaginal micronized progesterone will be administered at a total daily dose of 400 mg, given as Utrogestan® 200 mg (Besins Healthcare, France) twice daily, in the morning and at bedtime, from after randomization to 37+0/7 week of gestation or in case of preterm birth whatever comes first.

In both group, participants will be asked to record their vaginal progesterone application in a patient diary sheet for up to 140 days. At every visit, their compliance was documented by checking the diary and drug purchasing records from the hospital pharmacy. Compliance rate was calculated by dividing the number of progesterone doses used by the number of progesterone doses that should have been used since the last visit. Participants were considered compliant when their drugs used-to-prescribed rate was 80%.

Follow-up examination will be 7 days after randomization and then 2 weeks apart until delivery. At every exam, we perform routine antenatal care and CL measurement, record drug compliance and reveal any adverse events or complications. In case of premature rupture of the membranes, active vaginal bleeding, other signs of preterm labor, or severe discomfort of the participant, the use of cerclage and/or progesterone will be discontinued. Further treatment was indicated per local protocol. All interventions were terminated at 37 weeks or at delivery, whichever came first. Delivery will take place by either spontaneous onset of labor, induction of labor, or elective cesarean section according to national guidelines for twin pregnancies.

In cases where the patient delivers at hospitals that are not among the six study sites, data on neonatal and obstetric outcomes will be collected through telephone follow-up and medical record summaries obtained from the respective healthcare facilities.

The selected outcome measures correspond to the core outcome set established for studies on preterm birth prevention by GONet and the Core Outcomes in Women's Health initiative.

Hospital costs will be measured from hospital costs of patients and neonates.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18
* Twin pregnancy
* Asymptomatic short cervix (CL≤30mm) at routine ultrasound investigation
* Gestational age at 16+0- 24+0 weeks

Exclusion Criteria:

A potential paticipant who meets any of the following criteria will be excluded from participation in this trial:

* Women with twin pregnancy in which one or both fetuses are diagnosed with a major structural or congenital abnormality that is likely to influence the composite adverse neonatal outcome.
* Women with a monochorionic monoamniotic twin pregnancy
* A monochorionic twin pregnancy with twin-to-twin transfusion syndrome before or at the time of inclusion.
* Patients have indications for vaginal cerclage: Recurrent late miscarriage (from 14 weeks) or preterm birth occurring two or more times.
* Women with dilatation of the cervix diagnosed by ultrasound or physical exam
* Women with overt symptoms of preterm labor at the time of measurement of the short cervix (regular contractions, PPROM, recurrent blood loss).
* Women with the presence of fever ≥ 38 degrees Celsius.
* Women with a placenta previa, vasa previa.
* Uterine malformations: unicornuate uterus, bicornuate uterus, uterine septum, fibroid…
* Severe maternal conditions (heart failure, chronic kidney disease, systemic lupus erythematosus …)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be biologically female and pregnant
Enrollment: 260 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Preterm birth < 28 weeks | From randomization until 27 6/7 weeks
  Number of participants with preterm birth before 28 weeks of gestation

SECONDARY OUTCOMES:
Gestational age at birth | At birth
  Number of completed weeks and days of gestation at the time of delivery, calculated based on the date of embryo transfer for pregnancies conceived via in vitro fertilization (IVF), or by ultrasound measurement of the crown-rump length (CRL) of the larger fetus between 11 weeks and 13 weeks 6 days of gestation, or by head circumference measurement for pregnancies beyond 14 weeks of gestation.
Preterm birth < 32 weeks | From randomization until 31 6/7 weeks
  Number of participants with preterm birth before 32 weeks of gestation
Preterm birth < 34 weeks | From randomization until 33 6/7 weeks
  Number of participants with preterm birth before 34 weeks of gestation
Preterm birth < 37 weeks | From randomization until 36 6/7 weeks
  Number of participants with preterm birth before 37 weeks of gestation
Spontaneous preterm birth <28 weeks | From randomization until 27 6/7 weeks
  Number of participants with spontaneous preterm birth before 28 weeks of gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Spontaneous preterm birth < 32 weeks | From randomization until 31 6/7 weeks
  Number of participants with spontaneous preterm birth before 32 weeks of gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Spontaneous preterm birth < 34 weeks | From randomization until 33 6/7 weeks
  Number of participants with spontaneous preterm birth before 34 weeks of gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Spontaneous preterm birth < 37 weeks | From randomization until 36 6/7 weeks
  Number of participants with spontaneous preterm birth before 37 weeks of gestation, including preterm spontaneous rupture of membranes, preterm premature rupture of membranes (PPROM)
Iatrogenic preterm birth < 28 weeks | From randomization until 27 6/7 weeks
  Number of participants with non-spontaneously before 28 weeks of gestation
Iatrogenic preterm birth < 32 weeks | From randomization until 31 6/7 weeks
  Number of participants with non-spontaneously before 32 weeks of gestation
Iatrogenic preterm birth < 34 weeks | From randomization until 33 6/7 weeks
  Number of participants with non-spontaneously before 34 weeks of gestation
Iatrogenic preterm birth < 37 weeks | From randomization until 36 6/7 weeks
  Number of participants with non-spontaneously before 37 weeks of gestation
Preterm premature rupture of membranes | From randomization until delivery, assessed up to 37 weeks of gestation
  Number of participants diagnosed with preterm premature rupture of membranes (PPROM), defined as spontaneous rupture of membranes before 37 weeks of gestation and prior to the onset of labor. Diagnosis is based on clinical signs, including pooling of amniotic fluid in the vaginal vault.
Hospital costs | From randomization to the time of hospital discharge of both the mother and the neonate(s), assessed up to 90 days after delivery
  Total hospital-related cost per participant, including: Direct medical costs (e.g., fees for consultations, medications, antenatal and delivery monitoring, treatment of complications related to cervical cerclage, and neonatal care during hospitalization)
Maternal death | From randomization until maternal hospital discharge, assessed up to 28 days after delivery
  Death of the mother
Composite of maternal adverse outcome | From randomization until maternal hospital discharge, assessed up to assessed up to 28 days after delivery
  Number of participants who have any of the following maternal complications: chorioamnionitis, necrosis or rupture of the cervix, preterm premature rupture of the membranes, maternal death
Apgar score at 1 minute | Assessed at 1 minute after birth
  Apgar score at 1 minute
Apgar score at 5 minutes | Assessed at 5 minutes after birth
  Apgar score at 5 minutes
Apgar Score < 7 at 5 minutes | Assessed at 5 minutes after birth
  Apgar Score < 7 at 5 minutes
Birthweight | At birth
  The weight of the live-born infant measured in grams at birth
Number of neonates in need for respiratory supports | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates requiring respiratory support, including intubation, continuous positive airway pressure (CPAP), or high-flow nasal cannula (HFNC).
Length of ventilation | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of days the neonate required respiratory support with mechanical ventilation (invasive or non-invasive), counted from the initiation of ventilation until final discontinuation.
Respiratory distress syndrome | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates diagnosed with respiratory distress syndrome (RDS), based on clinical signs (chest movement, intercostal retraction, xiphoid retraction, nasal flaring, expiratory grunt) and classified by Silverman score.
Admission to the neonatal intensive care unit | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates admitted to the neonatal intensive care unit (NICU)
Length of neonatal intensive care unit stay | From admission to Neonatal Intensive Care Unit until neonatal hospital discharge or hospital referral, assessed up to 3 months corrected age
  Number of days of neonatal intensive care unit (NICU) stay
Length of neonatal admission | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Total number of days of neonatal hospitalization, including stays in the neonatal intensive care unit (NICU) and the neonatal department
Neonatal infection | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates with the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid (CSF), or catheterized/supra-pubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an X-ray confirming infection
Neonatal seizures | From delivery to neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates with neonatal seizures
Intra-ventricular hemorrhage grades III and IV | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates diagnosed with grade III or IV intraventricular hemorrhage by ultrasonography
Necrotizing enterocolitis (NEC) | From birth until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates diagnosed with necrotizing enterocolitis (NEC) based on the clinical signs triad of abdominal distension, gastrointestinal bleeding, and pneumatosis intestinalis (air in bowel wall on abdominal X-ray) classified by Modified Bell's criteria.
Neonatal sepsis | From birth until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates diagnosed with neonatal sepsis based on clinical signs (such as temperature instability, respiratory distress, lethargy, feeding difficulties) combined with laboratory evidence of infection (positive blood culture or other sterile site cultures) during the neonatal hospitalization period. The attending neonatologist confirms the diagnosis.
Neonatal referred hospital transfer for severe morbidities | From birth until referral to another neonatal hospital, assessed up to 3 months corrected age
  Number of neonates referred to other hospitals for severe morbidities
Stillbirth | From randomization until delivery, assessed up to assessed up to 28 days after delivery
  Number of participants with stillbirth occurring at or after 28 weeks of gestation during the study period.
Neonatal deaths | From birth until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of intrapartum, neonatal, and perinatal deaths
Composite neonatal adverse outcome | From birth until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates who have any of the following neonatal outcome: neonatal sepsis, respiratory distress syndrome, intraventricular hemorrhage grade III and IV, necrotizing enterocolitis, perinatal death.
Maternal side effects | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants with at least one of the following: chorioamnionitis, severe bleeding, cervical necrosis, or cervical rupture
Number of admission episodes for threatened preterm birth | From randomization until delivery, assessed up to 28 days after delivery
  Number of admission episodes for threatened preterm birth

OTHER OUTCOMES:
Number of patients with TTTS after randomization | From randomization until delivery, assessed up to 28 days after delivery
  Number of patients diagnosed with twin-to-twin transfusion syndrome (TTTS) after randomization
Number of participants diagnosed with TTTS after randomization who received treatment during the study period | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants diagnosed with TTTS after randomization who received fetoscopic laser photocoagulation, serial amnioreduction, septostomy, selective reduction, or expectant management, from diagnosis until delivery
Number of patients with preeclampsia | From randomization until delivery, assessed up to 28 days after delivery
  Number of patients diagnosed with preeclampsia
Number of participants diagnosed with gestational diabetes mellitus (GDM) who required insulin therapy during the study period | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants diagnosed with gestational diabetes mellitus (GDM) who required insulin therapy during the study period
Length of hospital stay for treatment of threatened preterm birth | From randomization until 36 6/7 weeks
  Cumulative duration of hospital stay for treatment of threatened preterm birth (days)
Number of participants diagnosed with congenital anomalies after randomization | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants diagnosed with congenital anomalies after randomization during the study period
Number of participants with rupture of the cervix during labor related to prior cerclage | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants with rupture of the cervix during labor related to prior cerclage
Number of participants diagnosed with chorioamnionitis | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants diagnosed with chorioamnionitis, defined as clinical intra-amniotic infection based on maternal fever (≥38.0°C) and at least two of the following criteria: uterine tenderness, fetal tachycardia (>160 beats per minute), maternal tachycardia (>100 beats per minute), foul-smelling amniotic fluid, or maternal leukocytosis (>15 × 10⁹/L).
Number of participants with vaginal delivery | From randomization until delivery, assessed up to 28 days after delivery
  Number of participants with vaginal delivery
Number of participants with maternal infection | From randomization until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants with fever (defined as a temperature ≥37.5 degrees Celsius), start of intravenous broad-spectrum antibiotics (with evidence of infection confirmed by clinical and subclinical presentation), endometritis, myometritis or urinary tract infection
Number of participants admitted to intensive care unit | From randomization until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants admitted to intensive care unit
Length of intensive care unit stay | From randomization until maternal hospital discharge, assessed up to 28 days after delivery
  Number of days in intensive care unit stay
Number of neonates requiring cardiopulmonary resuscitation (CPR) at birth | From delivery to 72 hours postnatal
  Defined as the number of live-born neonates who received cardiopulmonary resuscitation (CPR) immediately after birth, including interventions such as positive pressure ventilation, chest compressions, and/or administration of medications, as per neonatal resuscitation guidelines.
Reason for Neonatal Intensive Care Unit admission | From delivery until Neonatal Intensive Care Unit discharge, assessed up to 3 months corrected age
  Reason for Neonatal Intensive Care Unit admission such as: respiratory distress, hypoglycemia, seizures, etc
Length of neonatal hospital stay | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Total number of days from birth until hospital discharge for each live-born neonate.
Number of neonates with neonatal infection | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates with presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid (CSF), or catheterized/supra-pubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an X-ray confirming infection
Number of neonates with neonatal seizures | From delivery to neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates with neonatal seizures
Number of neonates with hypoglycemia | From delivery until neonatal hospital discharge, assessed up to 3 months corrected age
  Number of neonates with hypoglycemia
Number of neonates referred to other hospitals for severe morbidities | From delivery until neonatal hospital referral, assessed up to 3 months corrected age
  Number of neonates referred to other hospitals for severe morbidities
Number of participants with post-partum hemorrhage | Within 24 hours from delivery
  Defined as blood loss >500 ml at vaginal birth or >1000 ml at caesarean birth within 24 hours after birth
Number of participants having maternal post-partum blood transfusion | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants having maternal post-partum blood transfusion
Number of participants with uterine rupture | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants with uterine dehiscence (defined as clinically asymptomatic disruption of the uterus that is discovered incidentally at surgery) or rupture (defined as clinically significant rupture involving the full thickness of the uterine wall and requiring surgical repair)
Number of participants with hysterectomy | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Hysterectomy for any postpartum complications
Number of participants with other post-partum complications | From randomization until maternal hospital discharge, assessed up to 28 days after delivery
  Number of participants with at least one of the following: venous embolism, pulmonary embolism, stroke, or cardiac arrest
Number of participants referred to other hospital due to severe morbidities | From randomization until maternal hospital referral, assessed up to 28 days after delivery
  Number of participants referred to another hospital due to severe morbidities, including pulmonary embolism, stroke, and cardiorespiratory arrest.
Postpartum blood transfusion volume | From delivery until maternal hospital discharge, assessed up to 28 days after delivery
  Total volume of blood products (in milliliters) transfused to the participant after delivery, including packed red blood cells, whole blood, or other blood components, recorded from delivery until hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Anh D Nguyen, Prof, MD,PhD, Study Chair — National Hospital of Obstetrics and Gynecology
Locations (6):
- Vietnam (6):
  - Bac Ninh 1 Obstetrics and Pediatrics Hospital, Bac Ninh, Vietnam, Bắc Ninh
  - Bac Ninh 2 Obstetrics and Pediatrics Hospital, Bac Ninh, Vietnam, Bắc Ninh
  - National Hospital of Obstetrics and Gynecology, Hanoi
  - Hung Yen Obstetrics and Pediatrics Hospital, Hung Yen, Vietnam, Hưng Yên
  - Ninh Binh Obstetrics and Pediatrics Hospital, Ninh Binh, Vietnam, Ninh Bình
  - Quang Ninh Obstetrics and Pediatrics Hospital, Quang Ninh, Vietnam, Quang Ninh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akar B, Ceylan Y, Kahraman A, Kole E, Caliskan E. Centile charts of cervical length in singleton and twin pregnancies between 16 and 24 weeks of gestation. J Turk Ger Gynecol Assoc. 2023 Jun 7;24(2):114-119. doi: 10.4274/jtgga.galenos.2023.2022-7-3. Epub 2023 Mar 31. PMID 36999666
- [Result] He YTN, Pham HNH, Nguyen TC, Bui TQ, Vuong NT, Nguyen DTN, Le TV, Li W, Le CH, Ho TM, Mol BW, Dang VQ, Vuong LN. Cervical cerclage versus cervical pessary with or without vaginal progesterone for preterm birth prevention in twin pregnancies and a short cervix: A two-by-two factorial randomised clinical trial. PLoS Med. 2025 Feb 21;22(2):e1004526. doi: 10.1371/journal.pmed.1004526. eCollection 2025 Feb. PMID 39982935
- [Result] van 't Hooft J. A core outcome set for evaluation of interventions to prevent preterm birth: summary for CROWN. BJOG. 2016 Apr;123(5):666. doi: 10.1111/1471-0528.14003. No abstract available. PMID 27149346
- [Result] van 't Hooft J, Duffy JMN, Daly M, Williamson PR, Meher S, Thom E, Saade GR, Alfirevic Z, Mol BWJ, Khan KS; Global Obstetrics Network (GONet). A Core Outcome Set for Evaluation of Interventions to Prevent Preterm Birth. Obstet Gynecol. 2016 Jan;127(1):49-58. doi: 10.1097/AOG.0000000000001195. PMID 26646133
- [Result] D'Antonio F, Eltaweel N, Prasad S, Flacco ME, Manzoli L, Khalil A. Cervical cerclage for prevention of preterm birth and adverse perinatal outcome in twin pregnancies with short cervical length or cervical dilatation: A systematic review and meta-analysis. PLoS Med. 2023 Aug 3;20(8):e1004266. doi: 10.1371/journal.pmed.1004266. eCollection 2023 Aug. PMID 37535682
- [Result] Wu FT, Chen YY, Chen CP, Sun FJ, Chen CY. Outcomes of ultrasound-indicated cerclage in twin pregnancies with a short cervical length. Taiwan J Obstet Gynecol. 2020 Jul;59(4):508-513. doi: 10.1016/j.tjog.2020.05.007. PMID 32653121
- [Result] Freegard GD, Donadono V, Impey LWM. Emergency cervical cerclage in twin and singleton pregnancies with 0-mm cervical length or prolapsed membranes. Acta Obstet Gynecol Scand. 2021 Nov;100(11):2003-2008. doi: 10.1111/aogs.14255. Epub 2021 Sep 2. PMID 34476806
- [Result] Roman A, Zork N, Haeri S, Schoen CN, Saccone G, Colihan S, Zelig C, Gimovsky AC, Seligman NS, Zullo F, Berghella V. Physical examination-indicated cerclage in twin pregnancy: a randomized controlled trial. Am J Obstet Gynecol. 2020 Dec;223(6):902.e1-902.e11. doi: 10.1016/j.ajog.2020.06.047. Epub 2020 Jun 25. PMID 32592693
- [Result] Conde-Agudelo A, Romero R, Nicolaides K, Chaiworapongsa T, O'Brien JM, Cetingoz E, da Fonseca E, Creasy G, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone vs. cervical cerclage for the prevention of preterm birth in women with a sonographic short cervix, previous preterm birth, and singleton gestation: a systematic review and indirect comparison metaanalysis. Am J Obstet Gynecol. 2013 Jan;208(1):42.e1-42.e18. doi: 10.1016/j.ajog.2012.10.877. Epub 2012 Nov 15. PMID 23157855
- [Result] Jarde A, Lutsiv O, Park CK, Barrett J, Beyene J, Saito S, Dodd JM, Shah PS, Cook JL, Biringer AB, Giglia L, Han Z, Staub K, Mundle W, Vera C, Sabatino L, Liyanage SK, McDonald SD. Preterm birth prevention in twin pregnancies with progesterone, pessary, or cerclage: a systematic review and meta-analysis. BJOG. 2017 Jul;124(8):1163-1173. doi: 10.1111/1471-0528.14513. Epub 2017 Feb 8. PMID 28176485
- [Result] D'Antonio F, Berghella V, Di Mascio D, Saccone G, Sileo F, Flacco ME, Odibo AO, Liberati M, Manzoli L, Khalil A. Role of progesterone, cerclage and pessary in preventing preterm birth in twin pregnancies: A systematic review and network meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2021 Jun;261:166-177. doi: 10.1016/j.ejogrb.2021.04.023. Epub 2021 Apr 24. PMID 33946019
- [Result] Prediction and Prevention of Spontaneous Preterm Birth: ACOG Practice Bulletin, Number 234. Obstet Gynecol. 2021 Aug 1;138(2):e65-e90. doi: 10.1097/AOG.0000000000004479. PMID 34293771
- [Result] van Gils L, Dutilh R, Denswil N, Roman A, de Boer MA, Pajkrt E, Oudijk MA. The effectiveness of ultrasound-indicated cerclage for the reduction of extreme preterm birth in twin pregnancies with a short cervix: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2025 Jan;7(1):101555. doi: 10.1016/j.ajogmf.2024.101555. Epub 2024 Nov 26. PMID 39603526
- [Result] Khalil A, Sotiriadis A, Baschat A, Bhide A, Gratacos E, Hecher K, Lewi L, Salomon LJ, Thilaganathan B, Ville Y. ISUOG Practice Guidelines (updated): role of ultrasound in twin pregnancy. Ultrasound Obstet Gynecol. 2025 Feb;65(2):253-276. doi: 10.1002/uog.29166. Epub 2025 Jan 15. No abstract available. PMID 39815396
- [Result] Dang VQ, Nguyen LK, Pham TD, He YTN, Vu KN, Phan MTN, Le TQ, Le CH, Vuong LN, Mol BW. Pessary Compared With Vaginal Progesterone for the Prevention of Preterm Birth in Women With Twin Pregnancies and Cervical Length Less Than 38 mm: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):459-467. doi: 10.1097/AOG.0000000000003136. PMID 30741812
- [Result] Litwinska E, Syngelaki A, Cimpoca B, Frei L, Nicolaides KH. Outcome of twin pregnancy with two live fetuses at 11-13 weeks' gestation. Ultrasound Obstet Gynecol. 2020 Jan;55(1):32-38. doi: 10.1002/uog.21892. Epub 2019 Dec 13. PMID 31613412
- [Result] Osterman M, Hamilton B, Martin JA, Driscoll AK, Valenzuela CP. Births: Final Data for 2020. Natl Vital Stat Rep. 2021 Feb;70(17):1-50. PMID 35157571